CLINICAL TRIAL: NCT06954649
Title: Nutritional Intervention Study of the Effect of a Phytosterol-rich Extract on the Lipid Profile
Brief Title: Evaluation of the Functionality of an Extract Rich in Phytosterols and Phytostanols on Parameters Related to the Lipid Profile of Individuals With Hypercholesterolemia, Mainly in the Levels of Total Cholesterol, LDL Cholesterol and Oxidized LDL
Acronym: Hypolypox
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Centro de Edafología y Biología Aplicada del Segura (Other Government)
Collaborators: Universidad Católica San Antonio de Murcia (Other)
Responsible Party: Principal Investigator, Francisco A. Tomás-Barberán, Research Professor, Centro de Edafología y Biología Aplicada del Segura
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: CE102401; SNEO-20231059 (Other Grant/Funding Number: Ministry of Science, Innovation and Universities. Government of Spain)
Record Dates: First submitted 2025-04-24; First posted 2025-05-01 (Actual); Last update posted 2025-05-01 (Actual); Status verified 2025-04

CONDITIONS: Cholesterol Lowering; LDL Level
Keywords: cholesterol; LDL; HDL; oxidized LDL; triglycerides; phytosterols; bioactive compounds; resveratrol; hydroxytosol
MeSH Terms: interventions — Phytosterols; 3,4-dihydroxyphenylethanol

STUDY DESIGN:
Who Masked: Participant, Investigator
Masking Description: Clinical trial organizer (Universidad Católica San Antonio de Murcia, UCAM)
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Treatment group (Experimental): Experimental group. They will take an extract rich in phytosterols and phytostanols, resveratrol and hydroxytyrosol. They will take two capsules of the extract in the evening after dinner.
  Interventions: Dietary Supplement: Plant based extract rich in phytosterols and phytostanols resveratrol and hydroxytyrosol.
- Placebo group (Placebo Comparator): Control group. They will take a placebo supplement. They will take two capsules of the placebo, in the evening after dinner.
  Interventions: Other: Placebo

INTERVENTIONS:
Dietary Supplement: Plant based extract rich in phytosterols and phytostanols resveratrol and hydroxytyrosol. — Individuals will take two capsules daily of the phytosterol-rich extract for 56 days. Two capsules will be taken daily in the evening, after dinner
  Arms: Treatment group
Other: Placebo — Individuals will take two capsules daily of the placebo capsule for 56 days. Two capsules will be taken daily in the evening, after dinner
  Arms: Placebo group

SUMMARY:
The aim of this clinical trial is to evaluate the functionality of an extract rich in phytosterols and phytostanols on parameters related to the lipid profile of individuals with hypercholesterolemia, mainly on total cholesterol and LDL cholesterol levels

DETAILED DESCRIPTION:
A total of 45 participants with hypercholesterolemia (total cholesterol>200 mg/dL) will be recruited. Participants must not be taking any medication or nutritional supplement aimed at lowering cholesterol levels. Social networks and advertisements at the Universidad Católica San Antonio de Murcia (UCAM) and the Centro de Edafología y Biología Aplicada del Segura (CEBAS) will be used to recruit the individuals.

First, participants will attend to an informative session to learn in more detail about the objectives of the study and the procedures to be followed. In this session participants will sign the informed consent.

They will be divided into two groups:

* One group (n=23) that will take an extract rich in phytosterols and phytostanols (mainly β-sitosterol, β-sitostanol, campesterol and stigmasterol), resveratrol and hydroxytyrosol. The extract will be taken in capsule format.
* A control group (n=22) that will take a placebo supplement.

At the beginning of the study, anthropometric measurements of the participants will be taken. The participants' blood pressure will also be measured. An interview-questionnaire will be conducted to learn about and evaluate participants´s diet, physical activity and sleep quality. A blood sample will also be taken from the participants for biochemical analysis (total cholesterol, HDL, LDL, oxidized LDL, triglycerides and transaminases). From this day on, all participants will take two capsules daily of the phytosterol-rich extract or the placebo capsule, as appropriate, for 56 days. Capsules will be taken at night after dinner. Sampling and biochemical analysis will be repeated on days 28 and 56.

ELIGIBILITY:
Inclusion Criteria: total cholesterol>=200 mg/dl -

Exclusion Criteria: total cholesterol<200 mg/dl

-

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 45 (Actual)
Dates: Start 2025-01-14 (Actual); Primary Completion 2025-02-24 (Actual); Study Completion 2025-03-27 (Actual)

PRIMARY OUTCOMES:
Total cholesterol | From enrollment to the end of treatment at 56 days
  Change from baseline in total cholesterol levels measured at 28 and 56 days
Cholesterol LDL | From enrollment to the end of treatment at 56 days
  Change from baseline in cholesterol LDL levels measured at 28 and 56 days
Cholesterol HDL | From enrollment to the end of treatment at 56 days
  Change from baseline in cholesterol HDL levels measured at 28 and 56 days
Triglyceride | From enrollment to the end of treatment at 56 days
  Change from baseline in triglyceride levels measured at 28 days and 56 days
Transaminase | From enrollment to the end of treatment at 56 days
  Change from baseline in transaminase levels measured at 28 days and 56 days
Oxidized LDL | From enrollment to the end of treatment at 56 days
  Change from baseline in oxidized LDL levels measured at 28 and 56 days

CONTACTS AND LOCATIONS:
Locations (2):
- Spain (2):
  - Centro de Edafología y Biología Aplicada del Segura (CEBAS-CSIC), Murcia
  - Universidad Católica San Antonio de Murcia (UCAM), Murcia

IPD SHARING:
Plan to Share IPD: No